CLINICAL TRIAL: NCT07375212
Title: Acute Hemodynamic and Blood Volume Effects of Single-Dose Intranasal Bumetanide in Patients Implanted With the CardioMEMS™ and Cordella™ HF Systems: a 24-Hour Prospective Pilot Study
Brief Title: VAPorized Administration of Bumetanide for Outpatient Relief in Heart Failure
Acronym: VAPOR-HF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in Sponsor
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2341204
Record Dates: First submitted 2025-07-16; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure Congestive
Keywords: VAPOR-HF; Nasal Bumex; Nasal Bumetanide; Intranasal Bumex; Intranasal Bumetanide
MeSH Terms: conditions — Heart Failure | interventions — Bumetanide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intranasal Bumetanide Recipient (Other): All subjects in this study will receive the interventional drug, 4mg intranasal bumetanide,
  Interventions: Drug: Bumetanide, intranasal 4mg

INTERVENTIONS:
Drug: Bumetanide, intranasal 4mg — Intranasal route of administration for 4mg of bumetanide
  Other Names: Intranasal Bumex

SUMMARY:
This trial is seeking to determine whether a single 4mg intranasal dose of bumetanide acutely reduces pulmonary artery pressure and blood volume in the outpatient setting for patients with heart failure and an implanted device for remote patient monitoring (i.e. Cordella or CardioMEMS).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 y with chronic HF (NYHA II-III).
* Successful CardioMEMS or Cordella implantation ≥ 3 months prior.
* Clinically mild or worse congestion (no IV diuretics within 7 days).
* eGFR ≥ 20 mL/min/1.73 m²; serum K⁺ 3.5-5.2 mmol/L.

Exclusion Criteria:

* SBP < 90 mmHg, HR < 50 bpm, or > 110 bpm at baseline.
* Acute HF hospitalization < 30 days.
* Chronic nasal pathology or recent intranasal surgery.
* Known allergy to bumetanide or sulfamides.
* Pregnancy or lactation.
* Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device which has not reached its primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-21 (Actual); Primary Completion 2026-01-21 (Actual); Study Completion 2026-01-21 (Actual)

PRIMARY OUTCOMES:
Characterize Temporal Changes | 24 hours post-dose
  Characterize temporal changes in mean pulmonary artery pressure, systolic pulmonary artery pressure, diastolic pulmonary artery pressure, and heart rate at 1, 2, 3, 6, 12, and 24 hours post-dose of intranasal bumex.

SECONDARY OUTCOMES:
Quantify the Change in Total Blood Volume | 24 hours post-dose
  Quantify the change in total blood volume in milliliters 24 hours post-dose of intranasal bumex.
Changes in Pertinent Labs | 24 hours post-dose
  Describe the changes in the following labs at 24 hours post-dose of intranasal bumex: NT-proBNP, serum electrolytes, creatinine, hemoglobin, and hematocrit

CONTACTS AND LOCATIONS:
Overall Officials: Jason L Guichard, MD, PhD, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No